CLINICAL TRIAL: NCT03295227
Title: Feasibility Trial of Pembrolizumab in Unresectable Thymoma and Thymic Carcinoma
Brief Title: Pembrolizumab in Treating Participants With Unresectable Thymoma or Thymic Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0193; NCI-2018-01029 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0193 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-09-25; First posted 2017-09-27 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Stage III Thymoma AJCC v8; Stage IIIA Thymoma AJCC v8; Stage IIIB Thymoma AJCC v8; Stage IV Thymoma AJCC v8; Stage IVA Thymoma AJCC v8; Stage IVB Thymoma AJCC v8; Unresectable Thymic Carcinoma
MeSH Terms: conditions — Thymoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pembrolizumab) (Experimental): Participants receive pembrolizumab IV over 30 minutes on day 1. Courses repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase I trial studies the sides effects and best dose of pembrolizumab in treating participants with thymoma or thymic cancer that cannot be removed by surgery. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety/tolerability of pembrolizumab in unresectable patients with thymoma or thymic carcinoma who do not have pre-existing autoimmune diseases.

SECONDARY OBJECTIVES:

I. To evaluate the anti-tumor activity (response rate) of pembrolizumab in patients with unresectable thymoma or thymic carcinoma.

II. To evaluate the progression-free survival (PFS) and overall survival (OS) of pembrolizumab in patients with unresectable thymoma or thymic carcinoma.

EXPLORATORY OBJECTIVES:

I. We will test archival or fresh tumor tissue for PD-L1 immunohistochemistry (IHC).

II. We will perform Guardant360 blood analysis on patients with thymoma and thymic carcinoma to determine if any particular genetic mutations correlate to toxicities or clinical outcomes to pembrolizumab.

OUTLINE: This is a dose-escalation study.

Participants receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Courses repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up every 6 weeks for 1 year and then every 3 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable thymoma or thymic carcinoma.
* Any line of prior therapy allowed.
* Be willing and able to provide written informed consent/assent for the trial.
* Have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on day 1. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen.
* Have a performance status (PS) of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) PS.
* No history of or current diagnosis of a 'significant autoimmune disease" or paraneoplastic autoimmune disease, i.e. myasthenia gravis, Lambert-Eaton, systemic lupus, rheumatoid arthritis. For minor 'autoimmune' disorders such as psoriasis, arthritis (not including rheumatoid arthritis), Raynaud's disease; these are allowed onto trial.
* No active hepatitis or diagnosis of human immunodeficiency virus (HIV) disease.
* No prior malignancy unless it was cured over 2 years ago; i.e. prostate cancer, or early stage (I-III) solid tumors. Patients with a prior basal skin cancer or squamous cell carcinoma of the skin or in situ cervical malignancy that have undergone curative treatment are excluded from this requirement.
* Absolute neutrophil count >= 1500/mcL (within 10 days of treatment initiation).
* Platelets >= 100000mcL (within 10 days of treatment initiation).
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment) (within 10 days of treatment initiation).
* Serum creatinine OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) =< 1.5 X upper limit of normal (ULN) OR >= 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN (within 10 days of treatment initiation). Note: Creatinine clearance should be calculated per institutional standard.
* Serum total bilirubin =< 1.5 X ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN (within 10 days of treatment initiation).
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X ULN OR =< 5 X ULN for subjects with liver metastases (within 10 days of treatment initiation).
* Albumin >= 2.5 mg/dL (within 10 days of treatment initiation).
* International normalized ratio (INR) or prothrombin time (PT) activated partial thromboplastin time (aPTT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants (within 10 days of treatment initiation).
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential must be willing to use an adequate method of contraception, for the course of the study through 120 days after the last dose of study medication. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
* Male subjects of childbearing potential must agree to use an adequate method of contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has a known history of active TB (Bacillus tuberculosis).
* Hypersensitivity to pembrolizumab or any of its excipients.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent. - Note: Subjects with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study. - Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has a history of (non-infectious) pneumonitis that required steroids, or current pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies).
* Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus (HCV) ribonucleic acid (RNA) [qualitative] is detected).
* Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2017-12-06 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 3 years
  Frequency tables will be used to summarize categorical variables such toxicity type and severity.

SECONDARY OUTCOMES:
Progression-free survival | Up to 3 years
  Assessed by immune related Response Criterion (irRC) and immune-modified Response Evaluation Criteria in Solid Tumors (iRECIST). Kaplan-Meier estimates will be constructed. Confidence intervals around the median will be calculated using the Brookmeyer-Crowley method, confidence intervals around landmark time points will use the Greenwood formula for standard errors.
Overall survival assessed by iRECIST | Up to 3 years
  Kaplan-Meier estimates will be constructed. Confidence intervals around the median will be calculated using the Brookmeyer-Crowley method, confidence intervals around landmark time points will use the Greenwood formula for standard errors.
Overall response rate | Up to 3 years
  Assessed by RECIST 1.1 and iRECIST. Response rate and its 95% confidence interval will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Anne S Tsao, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org